CLINICAL TRIAL: NCT00486980
Title: A PHASE 3 MULTICENTER, RANDOMIZED, DOUBLE BLIND, PLACEBO-CONTROLLED STUDY TO EVALUATE THE EFFICACY AND SAFETY OF INTRAMUSCULAR PERAMIVIR IN SUBJECTS WITH UNCOMPLICATED ACUTE INFLUENZA
Brief Title: Intramuscular Peramivir for the Treatment of Uncomplicated Influenza
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was withdrawn for administrative reasons. The dose ranging plan for the program was revised".
Sponsor: BioCryst Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: BCX1812-312
Record Dates: First submitted 2007-06-14; First posted 2007-06-15 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2008-01

CONDITIONS: Influenza
Keywords: influenza
MeSH Terms: conditions — Influenza, Human | interventions — peramivir

INTERVENTIONS:
Drug: Peramivir 150mg
Drug: Peramivir 300mg

SUMMARY:
This is a multinational, randomized, double-blind study comparing the efficacy and safety of two single dose regimens of peramivir administered intramuscularly versus placebo in adults with uncomplicated acute influenza.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female subjects age ≥18 years
* A Rapid Antigen Test (RAT) performed on an adequate specimen collected from an anterior nasal swab. A negative initial RAT may be repeated within one hour of obtaining a negative result.
* Presence of fever at time of screening of ≥38.0 ºC (≥100.4 ºF) taken orally, or ≥38.5 ºC (≥101.2 ºF) taken rectally. For subjects with a positive RAT at the time of screening, a subject self-report of a history of fever or feverishness within the 24 hours prior to screening will also qualify for enrollment in the absence of documented fever at time of screening. For subjects with no positive RAT at screening, fever as defined above must be documented at time of screening
* Presence of at least one respiratory symptom (cough, sore throat, or nasal symptoms) of any severity (mild, moderate, or severe)
* Presence of at least one constitutional symptom (myalgia [muscle aches], headache, feverishness, or fatigue) of any severity (mild, moderate, or severe)
* Onset of symptoms no more than 48 hours before presentation for screening
* Written informed consent

Exclusion Criteria:

* Women who are pregnant or breast-feeding
* Presence of clinically significant signs of acute respiratory distress
* History of severe chronic obstructive pulmonary disease (COPD) or severe persistent asthma
* History of congestive heart failure requiring daily pharmacotherapy with symptoms consistent with New York Heart Association Class IV functional status within the past 12 months
* History of chronic renal impairment requiring hemodialysis and/or known or suspected to have moderate or severe renal impairment (actual or estimated creatinine clearance <50 mL/min)
* Current clinical evidence of active bacterial infection at any body site that requires therapy with oral or systemic antibiotics
* Presence of immunocompromised status due to chronic illness, previous organ transplant, or use of immunosuppressive medical therapy
* Current treatment for active viral hepatitis C
* Presence of known HIV infection with a CD4 count <350 cell/mm3
* Current therapy with oral warfarin or other systemic anticoagulant
* Receipt of any doses of rimantadine, amantadine, zanamivir, or oseltamivir in the 7 days prior to screening
* Immunized against influenza with live attenuated virus vaccine (FluMist®) in the previous 21 days
* History of alcohol abuse or drug addiction within 1 year prior to admission in the study
* Participation in a previous study of peramivir as treatment for acute influenza or previous participation in this study
* Participation in a study of any investigational drug within the last 30 days

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult